CLINICAL TRIAL: NCT07212595
Title: Biomarker and Renal Angina Validation to Assess Heart-Kidney Outcomes After Amino Acid Therapy
Acronym: BRAVE-HEART
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stuart Goldstein, MD (Other)
Collaborators: Congenital Heart Alliance of Cincinnati (Unknown)
Responsible Party: Sponsor-Investigator, Stuart Goldstein, MD, Professor of Pediatrics; Director, Center for Acute Care Nephrology, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 001 - BRAVE-HEART
Record Dates: First submitted 2025-09-28; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury; Mechanical Ventilation
Keywords: Cardiac Bypass; Pediatric; Acute Kidney Injury; Amino Acids
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acid Acid Infusion (Experimental): Amino Acid Infusion for up to 72 hours
  Interventions: Drug: Amino Acid infusion
- Placebo Infusion (Placebo Comparator): Placebo Infusion for up to 72 hours
  Interventions: Drug: Lactated ringers solution

INTERVENTIONS:
Drug: Amino Acid infusion — Amino acid infusion of 2 grams/kilogram of participant weight/day for up to 72 hours
  Other Names: Trophamine(TM) 10%
  Arms: Acid Acid Infusion
Drug: Lactated ringers solution — Placebo infusion to match the volume of the amino acid infusion in grams/kilogram/day
  Arms: Placebo Infusion

SUMMARY:
The goal of the BRAVE-HEART study is to learn if an amino acid infusion can reduce the risk of developing acute kidney injury after cardiac surgery in children. The main questions it aims to answer are:

1. Does an amino acid infusion decrease the number of participants with acute kidney injury?
2. Does an amino acid infusion decrease the number of days that participants are on a ventilator after cardiac surgery?

Researchers will compare amino acids to a placebo (a look-alike substance that contains no drug) to see if amino acids decrease the number of participants with acute kidney injury.

Participants will receive an amino acid or placebo infusion for up to 72 hours starting during cardiac surgery and only while in the operating room or the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Expected to be at high risk of developing acute kidney injury after cardiac surgery based on Age, The Society of Thoracic Surgeons-European Association for Cardio-Thoracic Surgery (STAT) score, and anticipated cardiopulmonary bypass time
* Age less than or equal to 18 years
* Weight greater than or equal to 5 kilograms

Exclusion Criteria:

* Preoperative extracorporeal organ support
* History of chronic kidney disease
* Known or suspected inborn errors of amino acid metabolism
* Known hypersensitivity to amino acids
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 3 times the upper limit of normal for age/gender
* Preterm infants less than 6 months of age who were born at less than 36 weeks gestational age
* Anuria at the time of randomization
* Expected use of total parental nutrition (TPN) within the first 72 hours post-operatively

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of acute kidney injury on post-operative days 2, 3, or 4 | From enrollment to post-operative day 4
  The rate of participants randomized to the amino acid infusion developing acute kidney injury as defined by Kidney Disease Improving Global Outcomes (KDIGO) as Stage 1, 2, or 3 will be compared to the rate of acute kidney injury in the placebo group
Rate of mechanical ventilation at 96 hours post-operatively | From enrollment to 96 hours post-operatively
  Rate of participants randomized to the amino acid infusion needing invasive mechanical ventilation beyond 96 hours post-operatively from congenital cardiac surgery repair will be compared to the rate from the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Goldstein, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
With a small data set from a single center, there is a high risk of the participants being able to be re-identified with the details within the data set.